CLINICAL TRIAL: NCT00139633
Title: Phase II Selective Dose Escalation of Chemoradiotherapy for Esophageal Cancer
Brief Title: Selective Dose Escalation for Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Oregon Clinic (Other)
Collaborators: Bristol-Myers Squibb (Industry); MedImmune LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETH097-02D
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2005-08-31 (Estimated); Status verified 2005-08

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer, chemotherapy, radiation
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Carboplatin; Fluorouracil; Paclitaxel; Radiation

INTERVENTIONS:
Drug: carboplatin, 5FU, Taxol and radiation

SUMMARY:
This prospective study was designed to assess the outcomes (survival and failure patterns) of therapy for localized esophageal cancer with conventional dose radiation (RT; 50.4 Gy) with concurrent continuous infusion 5-fluorouracil (5-FU) and weekly carboplatin/paclitaxel. Patients with less than complete response (CR) or partial response (PR) received dose escalation of radiation to 59.4 Gy with the same chemotherapy.

DETAILED DESCRIPTION:
we prospectively enrolled patients with T1-4, N0-1, M0-1a esophageal carcinoma to receive paclitaxel 45 mg/m2 IV over 1 hour and carboplatin AUC 2 IV over 30 minutes on days 1, 8, 15, 22, 29 and 36. 5-FU 225mg/m2 was delivered as a continuous infusion on days 1-38. RT was given 1.8Gy 5 days/wk for 5.5 wks (50.4Gy in 28 fx). After 6-8 weeks, patients underwent repeat staging with computed tomography (CT) scan, endoscopic ultrasound (EUS), and biopsy. Patients with a positive biopsy, or less than PR by CT and EUS, received a boost of 9 Gy with the same concurrent chemotherapy. Patients were followed every 4 months with CT/EUS first year, every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* T1-4, N0-1, M0-1a esophageal carcinoma

Exclusion Criteria:

* distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2000-07; Study Completion 2005-06

PRIMARY OUTCOMES:
survival at 4 years
local control at 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Seung, MDPhD, Study Chair — The Oregon Clinic
Locations (1):
- The Oregon Clinic, Portland, Oregon, United States